CLINICAL TRIAL: NCT03965741
Title: Prostate Cancer VTE in Sweden: Epidemiology and Anticoagulation Treatment of VTE
Brief Title: Study to Gather Information How Often Venous Thromboembolism Occurs in Prostate Cancer Patients in Sweden and How This Condition is Treated With Blood Thinners
Acronym: PRACTISE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20653
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; apixaban; Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men with Prostate Cancer (PCa)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Apixaban(Eliquis); Drug: Pradaxa (Dabigatran etexilate)
- Men without PCa

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Follow clinical administration
  Groups: Men with Prostate Cancer (PCa)
Drug: Apixaban(Eliquis) — Follow clinical administration
  Groups: Men with Prostate Cancer (PCa)
Drug: Pradaxa (Dabigatran etexilate) — Follow clinical administration
  Groups: Men with Prostate Cancer (PCa)

SUMMARY:
Patients with cancer are at a significantly increased risk of experiencing a venous thromboembolism (VTE). VTE is defined by a blood clot in the leg or lower extremity (deep vein thrombosis) or a blood clot in the lung (pulmonary embolism) and is a leading cause of condition of being diseased and death among cancer patients. The goal of the study is to gather information how often venous thromboembolism (VTE) occurs in prostate cancer patients in Sweden and how this condition is treated with blood thinners.

ELIGIBILITY:
Inclusion Criteria:

* Initially all patients newly diagnosed with PCa between 2007-2016 with at least one year before the end of follow up date (31 December 2017) will be included. From this population, a sub-population of PCa patients with a first cancer-related VTE event will be selected.

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Based on the data from the Prostate Cancer Database Sweden (PCBaSe), containing information from many national registries other than the Cancer register, such as Patient register, Dispensed drug register, Cause of Death registry and Population registries.
Sampling Method: Non-Probability Sample
Enrollment: 97765 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Subject's socio-demographic at the date of an incident PCa diagnosis | Retrospective analysis between 2007 and 2016
  Among men with PCa
Subject's clinical characteristics at the date of an incident PCa diagnosis | Retrospective analysis between 2007 and 2016
  Among men with PCa
Incidence rate of cancer-related VTE | Retrospective analysis between 2007 and 2016
  Among men with PCa
Cancer therapies in PCa at the initial time after diagnosis | Retrospective analysis between 2007 and 2016
  Among men with PCa
Choice of drug | Retrospective analysis between 2007 and 2016
  Among men with PCa and a first cancer-related VTE event； To characterize the long-term anticoagulation treatment
Duration of treatment | Retrospective analysis between 2007 and 2016
  Among men with PCa and a first cancer-related VTE event； To characterize the long-term anticoagulation treatment
Occurrence of recurrent VTE events | Retrospective analysis between 2007 and 2016
  Among men with PCa and a first cancer-related VTE event； By long-term anticoagulation treatment (LMWH (Low molecular weight heparin), VKA (Vitamin K anticoagulants) or NOAC (Non-vitamin K oral anticoagulation)) and its estimated duration (up 3 months, 3-6 months, more than 6 months)
Time between a first cancer-related and a recurrent VTE event | Retrospective analysis between 2007 and 2016
  Among men with PCa and a first cancer-related VTE event
Incidence rates of post-VTE bleeding events leading to hospitalization, and mortality by anticoagulation treatment | Retrospective analysis between 2007 and 2016
  Among men with PCa and a first cancer-related VTE event

SECONDARY OUTCOMES:
Subject's socio-demographic at the time of inclusion into the database | Retrospective analysis between 2007 and 2016
  Among PCa-free men from the general population
Subject's clinical characteristics at the time of inclusion into the database | Retrospective analysis between 2007 and 2016
  Among PCa-free men from the general population
Incidence rate of VTE events | Retrospective analysis between 2007 and 2016
  Among PCa-free men from the general population

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/